CLINICAL TRIAL: NCT05768997
Title: Prospective, Multicenter, Randomized Phase 3 Trial of High Dose IV Iron in Combination of Erythrocytosis Stimulating Agents in Chemotherapy Induced Anemia With Functional Iron Deficiency
Brief Title: High Dose IV Iron Plus ESA in Chemotherapy-induced Anemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, Zang, Dae Young, Principal Investigator, Hallym University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIGHEST-CIA
Record Dates: First submitted 2022-10-18; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — ferric derisomaltose; Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High dose IV iron plus ESA combination arm (Experimental)
  Interventions: Drug: Ferric Derisomaltose Injection; Drug: Darbepoetin Alfa Injection
- ESA monotherapy arm (Active Comparator)
  Interventions: Drug: Darbepoetin Alfa Injection

INTERVENTIONS:
Drug: Ferric Derisomaltose Injection — Ferric derisomaltose/iron isomaltoside (as iron) (0 weeks): 20mg/kg, diluted in 250ml of 0.9% physiological saline and injected intravenously over 30-60 minutes
  Arms: High dose IV iron plus ESA combination arm
Drug: Darbepoetin Alfa Injection — Darbepoietin alfa (0 weeks, 3 weeks, 6 weeks, 9 weeks): 6.75㎍/kg, subcutaneous or intravenous administration

SUMMARY:
This study is a multicenter, prospective, randomized phase 3 clinical study comparing the efficacy and safety of the combination treatment of ESA and high-dose IV iron (darbepoietin alfa + ferric derisomaltose/iron isomaltoside) with ESA monotherapy (darbepoietin alfa alone) in CIA patients with functional iron deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has signed a written consent

  * Age ≥ 19 ③ Histologically diagnosed advanced/metastatic solid cancer

    * Patients who have received myelosuppressive chemotherapy for palliative purposes within 1 month of participating in the study and plan to proceed with chemotherapy while participating in this study
    * Anemia with functional iron deficiency

      1. Hemoglobin <10g/dL
      2. functional iron deficiency: transferrin saturation <50% AND serum ferritin 30-800ng/mL ⑤ ECOG performance status 0-2 ⑥ life expectancy ≥ 24weeks

         Exclusion Criteria:
* Absolute iron deficiency (serum ferritin <30 ng/mL AND transferrin saturation <20%) or no iron deficiency (serum ferritin ≥800 ng/mL OR transferrin saturation ≥50%)

  * If there is another cause of anemia other than chemotherapy-induced anemia (eg, vitamin B12 or folic acid deficiency, hemolytic anemia, myelodysplastic syndrome, etc.)

    * Ongoing bleeding at the time of study registration

      * Patients who require rapid blood transfusion at the time of study registration (eg, rapidly progressing anemia)

        * Presence of bone marrow tumor invasion

          * Receiving erythropoiesis stimulating agents within 3 weeks of study registration or have a history of oral or intravenous iron administration or blood transfusion within 2 weeks of study registration

            * History of venous thromboembolism within 6 months or taking anticoagulants at the time of study registration

              * Past or family history of hemochromatosis ⑨ History of hypersensitivity to iron treatment or erythropoiesis stimulating agents ⑩ Uncontrolled acute or chronic infection ⑪ Renal dysfunction (serum creatinine ≥2.0 mg/dL, or glomerular filtration rate <30 mL/min/1.73 m2) or liver dysfuction (AST or ALT 3 times or more the upper limit of normal) ⑫ Pregnant or lactating women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean Hb change | from baseline to 12 weeks
  Mean change in Hb concentration from baseline to 12 weeks

SECONDARY OUTCOMES:
Hemoglobin response | during 12-week study period
  defined as an increase in Hb level of 2.0g/dL≥ from baseline value during 12-week study period
Time to hemoglobin response | during 12-week study period
Proportion of patients requiring RBC transfusion during 12-week study period | during 12-week study period
Quality of life assessment by Functional Assessment of Cancer Therapy-Anemia (FACT-An)/health-related quality of life instrument with 8 items (HINT-8)/EQ-5D-5L | during 12-week study period
Safety analysis | during 12-week study period
  Adverse events including AE of special interst (Anaphylaxis, Infusion reaction, Thromboembolic event)

CONTACTS AND LOCATIONS:
Locations (1):
- Hallym University Medical Center, Anyang-si, South Korea

IPD SHARING:
Plan to Share IPD: No